CLINICAL TRIAL: NCT01691599
Title: Infection Rates Following Internal Fixation of Open and Closed Tibia Fractures in India (INFINITI): a Prospective Multi-center Observational Study.
Brief Title: Infection Rates Following Internal Fixation of Open and Closed Tibia Fractures in India
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: INFINITI
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2015-06

CONDITIONS: Tibia Fracture
Keywords: Infection; Open tibia fractures; Closed tibia fractures; Wound infection
MeSH Terms: conditions — Tibial Fractures; Infections; Wound Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tibia fractures: Patients with open and closed tibia fracture treated with internal fixation in India

SUMMARY:
The objectives of this study are to investigate infection rates and management for open and closed tibia fracture subjects in India treated with internal fixation. These objectives will be carried out by answering the following questions:

1. What is the infection rate within one year of surgery for open and closed tibia fracture subjects in India treated with internal fixation?
2. What is the distribution of infection per type of infection, stratified by time (early, delayed, late) and location (superficial or deep) in open and closed tibia fracture subjects in India treated with internal fixation?

Secondary objectives

1. How are infections managed in open and closed tibia fracture subjects in India treated with internal fixation?
2. What is the treatment outcome for open and closed tibia fracture subjects in India treated with internal fixation?
3. What is the influence of the following clinic and subject factors on the occurrence of infection within one year for open and closed tibia fracture subjects in India treated with internal fixation?

   1. Hospital standard hygienic and antibiotic protocol for infection prevention
   2. Subject demographics
   3. Time between injury and surgery and between admission and surgery
   4. Fracture type (AO Müller classification)
   5. Soft tissue damage (according to the Tscherne classification for closed fractures or Gustilo classification for open fractures)
   6. Fracture management and implant type
   7. Surgical details such as duration of surgery
4. Is there a difference in health-related quality of life as measured by the EuroQol-5 Dimensions (EQ-5D) between subjects with and without infections?
5. Is there a difference in the number of complications not related to infection (adverse events and serious adverse events) between subjects with and without infections?

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who are 18 years of age or older.
2. Open or closed tibia fracture treated by internal fixation (plate or nail), or by external fixation with planned conversion to plate or nail.
3. Ability to understand the content of the subject information / informed consent form and to be willing to participate in the clinical investigation.
4. Written informed consent. Subjects with bilateral fractures will be included. In these subjects, the most severe fracture will be the one included in the study.

Exclusion Criteria:

1. Previous wound infection or osteomyelitis at the same limb (according to subject history).
2. Subjects who plan to undergo conversion surgery at a different hospital.
3. Previous fracture with retained hardware in injured extremity that will interfere with implant fixation.
4. Immunological deficiency disease.
5. Tumor related fractures.
6. Any severe systemic disease: class V-VI of the American Society of Anesthesiologists (ASA) physical status classification (Appendix 5).
7. Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment.
8. Subject is a prisoner.
9. Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with open or closed tibia fractures
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of infection | From surgery until the date of first documented infection assessed up to 1 year
  LAB (CRP + ESR level, Leukocyte count / diff.) and bacteriology of wound swabs / aspirated liquids and sensitivity testing, if the patient is suspected for a surgical site infection (SSI)

SECONDARY OUTCOMES:
Change in Quality of life measurement (EQ-5D) | Baseline and up to 5 day postoperative and 3months and 6months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prakash J Doshi, MD, Principal Investigator — Chief of Orthopaedics and Traumatology, Dr. Balabhai Nanavati Hospital, India
Locations (11):
- India (11):
  - Hi Tech Hospital, Gandhinagar, Gujarat
  - Dr. B.R. Ambedkar Medical College Hospital, Bangalore, Karnataka
  - MOSC Medical College, Kochi, Kerala
  - Kolhapur Institute of Orthopedics and Trauma, Kolhāpur, Maharashtra
  - Dr. Balabhai Nanavati Hospital, Mumbai, Maharashtra
  - Dr. R. N. Cooper Hospital, Mumbai, Maharashtra
  - Jai Hospital Pvt. Ltd., Nashik, Maharashtra
  - Sancheti Hospital, Pune, Maharashtra
  - Orthopedic Hospital and Post Graduate Institute of Swasthiyog Pratishthan, Sangli, Maharashtra
  - Post Graduate Institute of Medical Education and Research, Chandigarh, Punjab
  - Mukhopadhaya Orthopaedic Clinic and Research Centre, Bihār

REFERENCES:
- [Derived] Doshi P, Gopalan H, Sprague S, Pradhan C, Kulkarni S, Bhandari M. Incidence of infection following internal fixation of open and closed tibia fractures in India (INFINITI): a multi-centre observational cohort study. BMC Musculoskelet Disord. 2017 Apr 14;18(1):156. doi: 10.1186/s12891-017-1506-4. PMID 28410572